CLINICAL TRIAL: NCT00172497
Title: A Study of the Aggressive Acts Among Patients With Schizophrenia
Brief Title: Aggressive Acts Among Patients With Schizophrenia
Status: Suspended | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361700926
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2001-08

CONDITIONS: Schizophrenia
Keywords: aggressive acts
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this series of study has a many-fold intention depicted as follows: to describe and characterize schizophrenic patients' aggressive acts in hospital and community, to identify and specify heterogeneity in their structure, and to look for and set up risk factors for prevention. This study investigates four major issues: (1) Establishing an objective behavior rating scale for measuring aggressive acts; (2) Understanding the characteristics and incidence of aggressive acts by patients with schizophrenia; (3) Exploration of the heterogeneous structure of aggressive acts by patients with schizophrenia; and (4) Identifying the risk factors of aggressive acts of patients with schizophrenia.

DETAILED DESCRIPTION:
Psychiatric patients' aggressive acts can occur frequently and are recognized as a significant problem in psychiatric services. Understanding of aggressive acts in clinical settings and community is still incomplete and the clinical care of aggressive acts remains unsatisfactory. This study investigates four major issues: (1) Establishing an objective behavior rating scale for measuring aggressive acts; (2) Understanding the characteristics and incidence of aggressive acts by patients with schizophrenia; (3) Exploration of the heterogeneous structure of aggressive acts by patients with schizophrenia; and (4) Identifying the risk factors of aggressive acts of patients with schizophrenia. At first, the content validity, construct validity, and internal consistency of the Chinese version of Violence Scale were examined. Both of retrospective survey and prospective panel design were used for data collection. Patients fulfilling the DSM-IV criteria of schizophrenia in hospital and community, and their siblings and family caregivers, were recruited as different phases of study subjects, after signing informed consent for understanding their past history, prospective occurrence of aggressive acts, and the related risk factors. It is therefore to establish objective measures and to develop insights into the heterogeneity and related risk factors of aggressive acts, for improvement in the management and prevention of aggressive acts.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical diagnosis of schizophrenia spectrum, fulfilling the diagnostic criteria of the 4th version of Diagnostic and Statistical Manual (DSM-IV)(APA, 1994)were recruited as study subjects, after signing informed consent. Their families, including their siblings and family caregivers, were also recruited in the study.

Exclusion Criteria:

Exclusion criteria of the patient samples include co-mobility with mental retardation, personality disorder, organic brain disorders, and alcohol or substance abuse/ dependence.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2001-08; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Shing-Chia Chen, Ph.D., Principal Investigator — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan